CLINICAL TRIAL: NCT02777905
Title: Group Mindfulness-Based Cognitive Therapy for the Treatment of Late-Life Depression and Anxiety Symptoms in Primary Care: A Randomized Controlled Trial
Brief Title: Mindfulness-Based Cognitive Therapy for Depression and Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Dr. Karl Looper, Psychiatrist-in-Chief, Department of Psychiatry, Jewish General Hospital Co-Director, Mental Health Program, CIUSSS West-Central Montreal Health Associate Professor, Department of Psychiatry, McGill University, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-008
Record Dates: First submitted 2016-04-26; First posted 2016-05-19 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Symptoms of Depression; Symptoms of Anxiety
Keywords: late life; mindfulness meditation
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBCT intervention (Experimental): Mindfulness Based Cognitive therapy (MBCT) will consist of group meditative practices, lasting 2 hours per week (or whatever the patient can tolerate). The interventions will be conducted at the "centre local de services communautaires" (CLSC) Benny Farm, once a week. Patients will be invited to try various techniques during sessions. The patients will be encouraged to practice the Mindfulness techniques, that includes formal mindfulness meditation and informal mindfulness practices (e.g. being in the present moment while not meditating), at home, between sessions, and will be provided with meditation compact discs to help them do so. MBCT interventions also include a cognitive therapy perspective. Specifically, the interventionists will offer education regarding depression and anxiety and will work on automatic mental processes that are believed to be at the root of the recurrence of depressive and anxious symptoms.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Control Group (No Intervention): Patients randomized to the control group will be offered literature on mental health promotion and will receive treatment as usual in the primary care health center setting. After the end of the study, the control group will be offered MBCT.

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy
  Arms: MBCT intervention

SUMMARY:
About 10-20% of older patients in primary care suffer from symptoms of depression and/or anxiety. Depression and anxiety are associated with higher rates of cognitive decline, lower quality of life, increased medical comorbidity, and higher mortality rates in these patients. Given the world's aging population and consequent rapid increase in older patients in primary care, many traditional therapeutic approaches for depression or anxiety in this patient population - e.g. assessment by a mental health practitioner, individual psychotherapy and/or appropriate psychotropic medication - have been inadequate, with many patients having undetected depression and anxiety. Additionally, geriatric depression and anxiety are very common, but difficult to treat with psychotropic medications: patients are more sensitive to adverse effects and respond relatively less well to medication.

To help with this issue, the investigators are conducting a randomized controlled trial of mindfulness-based cognitive therapy (MBCT), a treatment that has been highly effective in treating depression and anxiety, but has not yet been assessed in older adults. There has been relatively little information about MBCT's effectiveness, particularly in the primary care setting and in the acute treatment of depression and anxiety(vs. maintenance treatment).

This study will be conducted in 75-100 older adults in primary care with symptoms of anxiety and depression. The study will take place in the "centre local de services communautaires" CLSC Benny Farm, a primary health care centre in Montreal, Canada. Most patients aged 60+ with symptoms of depression (Patient Health Questionnaire 9 (PHQ-9) score ≥10) or anxiety (General Anxiety Disorder-7 (GAD- 7) score ≥10) will be eligible. Patients who are eligible for the study will be randomized: half the patients will get 8-week MBCT with a trained interventionist (occupational therapist, psychiatry resident, or psychiatrist). The other half (control group) will get patient treatment as usual with patient primary care physician/primary care team during the study, but then after the study, patients will be offered the treatment if patients would like.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 60 years of age and above (clinical experience shows, that almost all patients with depressive and anxiety symptoms aged 60+ are able to participate in group MBCT)
* Patients with depression and/or anxiety symptoms as indicated by scores of ≥10 on the Patient Health Questionnaire (PHQ-9) and/or General Anxiety Disorder-7 (GAD- 7)
* Normal cognition or Mild Cognitive Impairment ("Normal" Result on the 3-minute Mini-Cog Test) [28]

Exclusion Criteria:

* Mild, Moderate, or Severe Dementia ("Abnormal" Result on the 3-minute Mini-Cog Test)
* Acute psychotic symptoms
* Severe personality problems that will interfere with their ability to function in a group setting
* Acute Suicidal ideation/intent
* Change in psychotropic medication during the 8 weeks of the intervention
* Hearing impairment not improved with hearing aids and/or sound amplification
* Unable to engage with MBCT for physical or practical reasons
* Ongoing Active Psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Significant decrease in the PHQ-9 (depression) score between baseline and 8-week follow-up | week 0 to 8 weeks
  Symptoms of depression will be assessed with the PHQ-9 at baseline and at at 8 weeks follow-up. Significant changes in these scores will be assessed after treatment.

SECONDARY OUTCOMES:
Decrease in the GAD-7 score (anxiety) between baseline and 8-week follow-up | week 0 to 8 weeks
  Symptoms of anxiety will be assessed with the GAD-7 questionnaire at baseline and at at 8 weeks follow-up. Significant changes in these scores will be assessed after treatment.

OTHER OUTCOMES:
Decreases in stress markers between baseline (week 0) and 8-week follow-up | week 0 to 8 weeks
  Blood draws will be performed to assess the levels of hypothalamus-pituitary-adrenal (HPA) axis activation and stress such as cortisol, dehydroepiandrosterone, adrenaline, noradrenaline and aldosterone. The concentrations will be given in pg/ml.
Decreases in inflammatory markers between baseline (week 0) and 8-week follow-up | week 0 to 8 weeks
  Blood draws will be performed to assess the levels of inflammatory markers such as C-reactive protein, cytokines, epidermal growth factor 1 (EGF-1) and indicators of the hypothalamus-pituitary-adrenal (HPA) axis activation and stress such as cortisol, dehydroepiandrosterone, adrenaline, noradrenaline and aldosterone. These measures will be taken at baseline and at 8-week follow-up. The concentrations will be given in pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- CLSC Benny Farm, Montreal, Quebec, Canada